CLINICAL TRIAL: NCT00653978
Title: Unilateral Versus Bilateral Stents for Bismuth Type II and III Malignant Hilar Strictures: A Prospective, Multi-center Randomized Controlled Trial
Brief Title: Unilateral Versus Bilateral Stents for Bismuth Type II and III Malignant Hilar Strictures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Zhaoshen Li, Changhai Hospital, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Changhai-080129
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2009-07

CONDITIONS: Cholangiocarcinoma
Keywords: ERCP; cholangiocarcinoma; hilar stricture
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patients receiving one stent
  Interventions: Procedure: ERCP plus one biliary stent
- 2 (Active Comparator): patients receiving two stents
  Interventions: Procedure: ERCP plus two biliary stents

INTERVENTIONS:
Procedure: ERCP plus one biliary stent — ERCP ＋ one biliary stent insertion
  Other Names: endoscopic retrograde cholangiopancreatography
  Arms: 1
Procedure: ERCP plus two biliary stents — ERCP ＋ two biliary stents insertion
  Other Names: endoscopic retrograde cholangiopancreatography
  Arms: 2

SUMMARY:
The aim of the present study was to compare the effect of unilateral versus bilateral stenting in patients with malignant hilar obstruction.

DETAILED DESCRIPTION:
Cholangiocarcinoma accounts for 3% of all gastrointestinal cancers and is the second commonest primary liver cancer. However only a few patients are suitable for surgical resection and therefore endoscopic biliary drainage is the most used palliative treatment modality for malignant hilar stricture. However, whether one or two stents can benefit the patients most is still to be defined. Numerous retrospective case series reached different conclusion, till now, only one randomized trial compared the effect of unilateral versus bilateral stenting in patients with malignant hilar obstruction, nonetheless, nearly one third of the patients had Bismuth Type I stricture, and one stent is enough for drainage in this situation, therefore, the best drainage strategy for patients with Bismuth Type II or Bismuth Type III malignant hilar obstruction is unknown. The aim of the present study was to compare the effect of unilateral versus bilateral stenting in patients with Bismuth Type II or III malignant hilar obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive untreated patients with biliary obstruction (Bismuth type II, III) at the hilum due to primary cholangiocarcinoma, gallbladder cancer, or periportal lymph node metastases. Diagnosis is based on US, CT, and MRCP.
* Histologic or cytologic confirmation of malignancy is established by percutaneous biopsy (US- or CT-guided) or by endoscopic tissue sampling, endoscopic brushing. Or the diagnosis is based on typical features on imaging and the expected clinical outcome during follow-up.
* All patients were considered unsuitable for resection on the basis of general medical condition and/or tumor extent.
* Full and informed consent is obtained.

Exclusion Criteria:

* Refuse to participate in this study.
* Refuse to provide informed consent.
* Refuse to be placed with plastic stents.
* Physically unfit for endoscopic treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Early complications | 30 days within treatment

SECONDARY OUTCOMES:
30-day mortality | 30 days within treatment
Late complications | 30 days after treatment
Median survival | From stent insertion to the death of the patient
Successful drainage | One month after stent insertion

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (2):
- Changhai Hospital, Second Military Medical University, Shanghai, China
- Department of Surgery and Transplant Center, Astrova, Slovakia